CLINICAL TRIAL: NCT05402826
Title: The Effect of Co-administration of Zinc and Vitamin E Oral Supplements on Short-term Postoperative Outcomes and Plasma Concentrations of Oxidative Stress Biomarkers in Cardiac Surgery Patients
Brief Title: Effect of Oral Zinc and Vitamin E Supplementation on Short-term Postoperative Outcomes in Cardiac Surgery Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Kerman University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 30285
Record Dates: First submitted 2022-05-21; First posted 2022-06-02 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Heart Surgery
MeSH Terms: interventions — Zinc; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive placebo pills.
  Interventions: Dietary Supplement: Placebo
- Zinc+vitamin E supplements (Active Comparator): Patients will receive zinc tablets plus alpha-tocopherol.
  Interventions: Dietary Supplement: Oral zinc + vitamin E

INTERVENTIONS:
Dietary Supplement: Oral zinc + vitamin E — In the zinc + vitamin E supplementation group, patients will receive a cumulative dose of 120 mg of oral zinc supplementation plus a cumulative dose of 1200 IU of oral vitamin E before surgery. After surgery, from the second day to the end of the hospital stay, patients receive 30 mg of zinc supplement plus 200 units of vitamin E per day.
  Arms: Zinc+vitamin E supplements
Dietary Supplement: Placebo — Patients in the placebo group will receive placebo pills before and after surgery.
  Arms: Placebo

SUMMARY:
Cardiac surgery can cause oxidative stress due to ischemia-reperfusion. Using antioxidants during perioperative period may help improve this condition. Vitamin E and zinc have antioxidant effects. In this study, the effects of oral co-administration of zinc and vitamin E supplements on short-term postoperative outcomes in cardiac surgery patients will be investigated.

DETAILED DESCRIPTION:
Cardiac surgery is a life-saving invasive procedure that may often be associated with significant postoperative complications. Cardiac surgery can cause oxidative stress due to ischemia-reperfusion. This is a post-ischemic complication that occurs when blood circulation is restored and causes inflammation and oxidative damage. Cardiac surgery with reperfusion injury can adversely affect the prognosis. Thus, reducing the extend of reperfusion injury and its associated pathways can be considered an important clinical issue. Reducing oxidative stress and inflammation may play an important role in the outcomes of heart surgery. Using antioxidants in pre or post surgery may help improve this condition. Vitamin E is a well-known fat-soluble antioxidant that prevents lipid peroxidation. Zinc has several roles including antioxidant effects. Zinc acts as a cofactor for important enzymes that contribute to the proper functioning of the antioxidant defense system. In addition, the mineral is involved in reducing free radicals by inducing metallothionein synthesis and circulating zinc concentration decreases significantly after surgery. In this study, the effects of oral co-administration of zinc and vitamin E supplements shortly before and after surgery on short-term postoperative outcomes, plasma concentrations of biomarkers of oxidative stress and inflammation in patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for open heart surgery (coronary artery bypass grafting)

Exclusion Criteria:

* Frequent use of multivitamin, zinc, vitamin E, vitamin C, omega-3 supplements over the past month
* Active cancer, chronic rheumatic disease, ESRD, liver cirrhosis, severe infection (WBC> 12000 mm3) before surgery
* Continued use of corticosteroids or NSAIDs for two weeks prior to admission (except A.S.A)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
ICU LOS | Through study completion, an average of 5 days
  Duration of patients' stay in the intensive care unit
Post surgery hospital LOS | Through study completion, an average of 10 days
  Duration of patients' stay in the hospital

SECONDARY OUTCOMES:
The sequential organ failure assessment score | On the third day after surgery
  Higher scores mean a worse outcome.
Plasma superoxide dismutase activity | up to 3 days after surgery
  Plasma superoxide dismutase activity in patients studied before surgery and three days after surgery
Plasma total antioxidant | up to 3 days after surgery
  Plasma total antioxidant capacity in patients studied before surgery and three days after surgery
Plasma CRP | up to 3 days after surgery
  Plasma C-reactive protein level in patients studied before surgery and three days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shafa Hospital, Kerman University of Medical Sciences, Kerman, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makiabadi E, Nakhaeizadeh R, Soleimani M, Nasrollahzadeh J. Effects of perioperative vitamin E and zinc co-supplementation on systemic inflammation and length of stay following coronary artery bypass graft surgery: a randomized controlled trial. Eur J Clin Nutr. 2024 Feb;78(2):120-127. doi: 10.1038/s41430-023-01356-x. Epub 2023 Oct 27. PMID 37891226